CLINICAL TRIAL: NCT05225818
Title: Preparing Successful Aging Through Dementia Literacy Education And Navigation (PLAN)-Home Pilot
Brief Title: Preparing Successful Aging Through Dementia Literacy Education And Navigation (PLAN)-Home
Acronym: PLAN-Home
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Our study design changed
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00299252
Record Dates: First submitted 2022-01-24; First posted 2022-02-07 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Dementia
Keywords: Nurse Practitioners; Diagnosis; Social Support; Patient Education
MeSH Terms: conditions — Dementia; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: PLAN - Home (Experimental): Trained NPs will deliver the PLAN-Home to the enrolled participants, which consists of home-based dementia evaluation, education, and care planning for older adults with probable dementia.
  Interventions: Behavioral: PLAN - Home
- No intervention: Control Group (No Intervention): The control group will receive a copy of the publicly available educational material on 10 warning signs and symptoms of Alzheimer's disease and action steps prepared by Alzheimer's Association.

INTERVENTIONS:
Behavioral: PLAN - Home — home-based intervention program for dementia evaluation, education, and care planning
  Arms: Experimental: PLAN - Home

SUMMARY:
Rapid growth in elderly population and higher prevalence of dementia necessitates further attention to dementia. Even though early detection and continuing care are mainstays of dementia care, limited access to dementia diagnosis and dementia care planning for elders could be attributed to factors like low dementia literacy-the capacity to obtain, process, and understand basic dementia-related information and services to make appropriate health decisions-and lack of social support. Developing innovative pathways to transition families of individuals with probable dementia into healthcare access for early diagnosis of dementia and timely dementia care planning can benefit patients and the patients' families. To this end, the investigators' study aims are to develop a home-based intervention program for dementia evaluation, education, and care planning and test its feasibility and acceptability in a pilot study.

DETAILED DESCRIPTION:
This research is being done to understand how an education and navigation support program led by trained Nurse Practitioners (NPs) helps older adults with probable dementia and the patients' caregivers. In a 2-arm randomized controlled trial (RCT) with 40 dyads, the investigators' aims are to (1) test the effect of a community-based intervention delivered by trained NPs for undiagnosed older adults with probable dementia and the patients' caregivers, (2) evaluate the effect of the PLAN on improving caregiver's dementia literacy, self-efficacy in dementia care and service use, social support, depression, and quality of life at 6 months in comparison to a group of participants who receive a copy of the publicly available educational material, and (3) examine whether the effect of PLAN differs across age, sex, and education caregiver subgroups.

Aim 1 tests the following hypotheses: older adults with probable dementia who receive the PLAN will have higher rates of linkage to medical service for dementia than those in the control group. Aim 2 tests the following hypothesis: caregivers in the PLAN group will have higher dementia literacy, self-efficacy in dementia care and service use, social support, and quality of life, and lower depression than those in the control group.

ELIGIBILITY:
Inclusion Criteria (Patient):

* Age 65 years or older
* Enrolled in home-based primary care
* Mini-Mental State Exam (MMSE) <24
* Has a caregiver who lives in the same household or has at least weekly interactions
* Able to consent or has a proxy available for consent
* Written consent to participate in the study

Inclusion Criteria (Caregiver):

* Age 18 years or older
* Able to read, write, and speak English
* Lives in the same household with an older adult with MMSE <24 or has at least weekly interactions
* Written consent to participate in the study

Exclusion Criteria (Patient):

* Previous dementia diagnosis
* All Axis I diagnoses other than depressive disorders (e.g., schizophrenia, bipolar disorder, or substance use disorder)
* Neurological disorders other than Alzheimer's disease that might affect cognition (e.g., stroke)
* Use of psychotropic drugs including antipsychotics

Exclusion Criteria (Caregiver):

* Plan to move from the area within 6 months
* Active treatment for a terminal illness or in hospice

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants linked to medical service for dementia | 6 months
  Number of participants linked to medical service for dementia measured by medical record verification. Linkage to medical service for dementia is defined as having had primary care or specialty care provider evaluation for cognitive impairment.

SECONDARY OUTCOMES:
Number of participants who complete a plan for dementia care | 6 months
  Completion of a plan for dementia care is measured by study questionnaire: "yes" or "no".
Number of participants who complete advanced directives | 6 months
  Completion of advanced directives is measured by study questionnaire: "yes" or "no".
Change in functional ability for activities of daily living as assessed by Katz scores | Baseline and 6 months
  The Katz Index of Independence in Activities of Daily Living is a 7-item instrument, with 1 point assigned for each item respondents are able to perform independently without supervision, direction, or guidance. Scores range from 0 to 6 with higher scores indicating higher independence.
Change in functional ability for instrumental activities of daily living as assessed by Lawton-Brody scores | Baseline and 6 months
  The Lawton-Brody Instrumental Activities of Daily Living Scale is an 8-domain instrument (5 domains historically used for men), with 1 point assigned for each statement that reflects higher levels of functioning. Summary scores range from 0 to 8 (5 for men) with higher scores indicating higher functioning and independence.
Change in Patient quality of life as assessed by Quality of Life-Patient scores (for all patient participants) | Baseline and 6 months
  QoL-dementia older adult is a 13-item instrument and scoring ranges from "poor" coded as 1 to "excellent" coded as 4 for each item. Total scores will range from 13 to 52 with higher scores indicating higher quality of life.
Change in Dementia Literacy as assessed by Rapid Estimate of Adult Literacy in Medicine (REALM)-Dementia scores (for all caregiver participants) | Baseline and 6 months
  The dementia literacy test is a 11-item instrument. Scoring of the dementia literacy instrument is in such a way that each correct response will be coded as 1 whereas incorrect response will be coded as 0. Total scores can range from 0 to 11 with higher scores indicating higher dementia literacy.
Change in Social Support as assessed by Medical Outcomes Study (MOS)-Social Support survey scores (for all caregiver participants) | Baseline and 6 months
  The 8-item scale of medical outcomes study scoring ranges from "none of the time" coded as 1 to "all of the time" coded as 5 for each item. Total scores will range from 8 to 40 with higher scores indicating higher social support.
Change in depression as assessed by Patient Health Questionnaire-2 (for all caregiver participants) | Baseline and 6 months
  Patient health questionnaire-2 is a 2-item instrument and scoring ranges from "not at all" coded as 0 to "nearly every day" coded as 3. Total scores will range from 0 to 6 with higher score indicating greater depressive symptoms.
Change in self-efficacy as assessed by Self-Efficacy Dementia Scale scores | Baseline and 6 months
  Dementia self-efficacy scale is a 10-item instrument. Scoring of the dementia self-efficacy scale ranges from "not at all certain" coded as 1 to "very certain" coded as 10 for each item. Total scores will range from 10 to 100 with higher scores indicating higher self-efficacy.
Change in Caregiver Quality of Life | Baseline and 6 months
  QoL-dementia caregiver is a 13-item instrument and scoring ranges from "poor" coded as 1 to "excellent" coded as 4 for each item. Total scores will range from 13 to 52 with higher scores indicating higher quality of life.
Program satisfaction as assessed by study questionnaire | 6 months
  Caregiver satisfaction with the intervention program will be measured on a 10-point visual analogue scale, with scoring ranges from 0 "not at all satisfied" to 10 "extremely/highly satisfied". Higher scores will indicate greater satisfaction with program.

CONTACTS AND LOCATIONS:
Overall Officials: Haera Han, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson L, Tang E, Taylor JP. Dementia: timely diagnosis and early intervention. BMJ. 2015 Jun 16;350:h3029. doi: 10.1136/bmj.h3029. No abstract available. PMID 26079686
- [Background] Landers S, Madigan E, Leff B, Rosati RJ, McCann BA, Hornbake R, MacMillan R, Jones K, Bowles K, Dowding D, Lee T, Moorhead T, Rodriguez S, Breese E. The Future of Home Health Care: A Strategic Framework for Optimizing Value. Home Health Care Manag Pract. 2016 Nov;28(4):262-278. doi: 10.1177/1084822316666368. Epub 2016 Oct 5. PMID 27746670
- [Background] Vespa J. (March 13, 2018). The graying of America: More older adults than kids by 2035. United States Census Bureau. Retrieved from https://www.census.gov/library/stories/2018/03/graying-america.html.
- [Background] Centers for Medicare & Medicaid Services. (February 06, 2019). New app displays what original Medicare covers. Retrieved from https://www.cms.gov/newsroom/press-releases/new-app-displays-what-original-medicare-covers#:~:text=The%20Medicare%20population%20is%20projected,almost%20daily%20(65%20percent).
- [Background] Yao NA, Rose K, LeBaron V, Camacho F, Boling P. Increasing Role of Nurse Practitioners in House Call Programs. J Am Geriatr Soc. 2017 Apr;65(4):847-852. doi: 10.1111/jgs.14698. Epub 2016 Dec 28. PMID 28029709
- [Background] Keenan TA. (November 2010). Home and community preferences of the 45+ population. AARP Research. Retrieved from http://www.aarp.org/research/topics/community/info-2014/home-community-services-10.html.
- [Background] Ng T, Harrington C, Musumeci M, Reaves EL. (November 3, 2015). Medicaid home and community-based services programs: 2012 data update. Kaiser Family Foundation. https://www.kff.org/medicaid/report/medicaid-home-and-community-based-services-programs-2012-data-update/.
- [Background] Prasad S, Dunn W, Hillier LM, McAiney CA, Warren R, Rutherford P. Rural geriatric glue: a nurse practitioner-led model of care for enhancing primary care for frail older adults within an ecosystem approach. J Am Geriatr Soc. 2014 Sep;62(9):1772-80. doi: 10.1111/jgs.12982. PMID 25243682
- [Background] Jaffe S. Home Health Care Providers Struggle With State Laws And Medicare Rules As Demand Rises. Health Aff (Millwood). 2019 Jun;38(6):981-986. doi: 10.1377/hlthaff.2019.00529. No abstract available. PMID 31158027
- [Background] Maryland Health Care Commission. Home Health Utilization Tables and Agency Data Collection. Table 13: Total Number of Clients (Unduplicated Count) by Jurisdiction of Residence, Payment Source and Agency, Fiscal Year 2008. 2020 [cited 2021 November 19]. Available from https://mhcc.maryland.gov/public_use_files/index.aspx.
- [Background] Maryland Health Care Commission. Home Health Utilization Tables and Agency Data Collection. Table 13: Total Number of Clients (Unduplicated Count) by Jurisdiction of Residence, Payment Source and Agency, Fiscal Year 2018. 2020 [cited 2021 November 19]. Available from https://mhcc.maryland.gov/public_use_files/index.aspx.
- [Background] Osakwe ZT, Aliyu S, Sosina OA, Poghosyan L. The outcomes of nurse practitioner (NP)-Provided home visits: A systematic review. Geriatr Nurs. 2020 Nov-Dec;41(6):962-969. doi: 10.1016/j.gerinurse.2020.07.001. Epub 2020 Jul 24. PMID 32718756
- [Background] Wolff-Baker D, Ordona RB. The Expanding Role of Nurse Practitioners in Home-Based Primary Care: Opportunities and Challenges. J Gerontol Nurs. 2019 Jun 1;45(6):9-14. doi: 10.3928/00989134-20190422-01. PMID 31135933
- [Background] Echeverry LM, Lamb KV, Miller J. Impact of APN Home Visits in Reducing Healthcare Costs and Improving Function in Homebound Heart Failure. Home Healthc Now. 2015 Nov-Dec;33(10):532-7. doi: 10.1097/NHH.0000000000000304. PMID 26529444
- [Background] Coppa D, Winchester SB, Roberts MB. Home-based nurse practitioners demonstrate reductions in rehospitalizations and emergency department visits in a clinically complex patient population through an academic-clinical partnership. J Am Assoc Nurse Pract. 2018 Jun;30(6):335-343. doi: 10.1097/JXX.0000000000000060. PMID 29878967
- [Background] Smits M, Peters Y, Ranke S, Plat E, Laurant M, Giesen P. Substitution of general practitioners by nurse practitioners in out-of-hours primary care home visits: A quasi-experimental study. Int J Nurs Stud. 2020 Apr;104:103445. doi: 10.1016/j.ijnurstu.2019.103445. Epub 2019 Sep 28. PMID 32105972
- [Background] Medicare.gov. (n.d.). Home health services. Retrieved from https://www.medicare.gov/coverage/home-health-services.
- [Background] Dobson DaVanzo & Associates. (2014, March 25). Updated report: Impact of proposed legislation H.R. 2504/S. 1332 on Medicare expenditures [memorandum]. Retrieved from http://www.nahc.org/assets/1/7/Dobson_DaVanzo_Impact_Memo_Revised_3_25_14.pdf.
- [Background] US Congress. (2019). S.296-Home Health Care Planning Improvement Act of 2019. Retrieved from https://www.congress.gov/bill/116th-congress/senate-bill/296.
- [Background] Mora K, Dorrejo XM, Carreon KM, Butt S. Nurse practitioner-led transitional care interventions: An integrative review. J Am Assoc Nurse Pract. 2017 Dec;29(12):773-790. doi: 10.1002/2327-6924.12509. Epub 2017 Aug 28. PMID 28845555